CLINICAL TRIAL: NCT00595491
Title: Inflammatory Cellular Trafficking in Asthma in Response to Segmental Allergen Challenge
Brief Title: Pilot Study to Identify the Mediators and Inflammatory Cell Surface Receptors Involved in Allergic Airway Inflammation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benjamin Medoff (Other)
Collaborators: National Institutes of Health (NIH) (NIH); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Benjamin Medoff, Chief, Pulmonary and Critical Care Unit, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007-P-001050; NIH 4 R37 AI040618 (Other: NIH); BB-IND 13094 (Other: FDA); W81XWH-16-1-0493 (Other Grant/Funding Number: U.S. Army Medical Research)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Asthma; Inflammation; Allergic; Airway; Challenge; Chemokines
MeSH Terms: conditions — Asthma; Inflammation | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- allergic asthmatic, allergic nonasthmatic, healthy (Experimental): Adults who are allergic asthmatics, allergic nonasthmatics, or healthy controls will receive segmental allergen challenge to the lung
  Interventions: Biological: Bronchoscopy, Segmental Allergen Challenge, and Broncheoalveolar Lavage

INTERVENTIONS:
Biological: Bronchoscopy, Segmental Allergen Challenge, and Broncheoalveolar Lavage — Bronchoalveolar lavage is performed in the lingula without instillation of diluent or allergen. A 2ml aliquot of diluent is instilled into the right upper lobe. The procedure is repeated in the right middle lobe with instillation of 2ml of Cat or Mite allergen. A test dose of allergen is administered first. This will consist of 2ml allergen at 1/10th the threshold concentration for Cat or DF Mite Allergen or at 1/30th the threshold concentration for DP Mite Allergen. If on visual inspection through the bronchoscope there is no evidence of reaction to the test dose, a 2nd allergen challenge is done in the right middle lobe using 2ml of full-dose allergen. After a 1,6, or 24hr recovery period, a single 2nd bronchoscopy is performed after delivery of allergen extract and diluent and 1 Tbsp of blood is obtained. Bronchoalveolar lavage will be obtained from the lobes in which the diluent and allergen were instilled. OFDI and endobronchial brushing of the airways will also be performed.
  Other Names: One of 3 Standardized allergen extracts will be used:; Standardized Cat Hair Extract; Standardized mite extract-Dermatophagoides farinae; Standardized mite extract-Dermatophagoides pteronyssinus; Phenolized saline diluent will also be used in this study.; All will be purchased from Greer Laboratories Lenoir,NC.

SUMMARY:
Asthma is a heterogeneous disorder in which multiple potential inflammatory pathways contribute to airway obstruction. The biological basis for airway inflammation is the subject of intensive investigation. This work is designed to identify airway factors that are responsible for recruiting cells and associate their airway presence with atopy and asthma.

DETAILED DESCRIPTION:
The production of chemotactic cytokines or chemokines by the airways is one of the mechanisms thought to be responsible for the recruitment of inflammatory cells to the airways (Makay 2001). While the chemokine receptor-ligand systems responsible for immune cell homing to the mucosal surface of the gastrointestinal tract have been clarified, those responsible for allergic airway inflammation remain unknown. This work is designed to identify airway factors that are responsible for recruiting cells and associate their airway presence with atopy and asthma.

ELIGIBILITY:
A. Subjects with Allergic Asthma (AA subjects)

Inclusion Criteria:

1. All subjects will have a baseline FEV1 determined at the characterization visit that is no less than 75 % of the predicted value.
2. All subjects will have a clinical history of allergic symptoms to cat or dust mite allergen and demonstrated skin reactivity (a positive allergen prick test).
3. Life-long absence of cigarette smoking (defined as a lifetime total of less than 5 pack-years); none in 5 years).
4. Willing and able to give informed consent.
5. Expressed the desire to participate in an interview with the principal investigator.
6. Age between 18 and 50 years.

Exclusion Criteria:

1. Women of childbearing potential who are documented to be pregnant (based on Urine beta-HCG testing), are sexually active and not using contraception, are seeking to become pregnant, or who are nursing.
2. The presence of spontaneous asthmatic episode or clinical evidence of upper respiratory tract infection within the previous 6 weeks.
3. Participation in research study involving a drug or biologic during the 30 days prior to the study.
4. Intolerance to albuterol, atropine, lidocaine, fentanyl, or midazolam.
5. Antihistamines within 7 days of the screening visit.
6. Presence of diabetes mellitus, congestive heart failure, ventricular arrhythmias, history of a cerebrovascular accident, renal failure, history of anaphylaxis, or cirrhosis.
7. Use of systemic steroids, increased use of inhaled steroids, beta blockers and MAO inhibitors or a visit for an asthma exacerbation within 1 month of the screening visit.
8. Antibiotic use for respiratory disease within 1 month of the characterization visit or a respiratory tract infection within 6 weeks of the bronchoscopy visits.
9. A history of asthma-related respiratory failure requiring intubation.
10. Quantitative skin-prick test positive reaction down to an allergen concentration of 0.056 BAU or AU/ml .
11. Taking beta-adrenergic blocking agents or monoamine oxidase inhibitors.
12. Subjects with a high possibility of poor compliance with the study.
13. No history of cigarette smoking within the past 5 years or > 10 pack years total.
14. Having second-hand cigarette smoke exposure or indoor furry pets except in the case of dog, if the subject is not allergic to the dog and the subject has a negative skin test to dog (It is also preferred but not required that dust mite allergic subjects have dust mite-proof encasings on their mattress and pillows.)
15. Other lung diseases, such as sarcoidosis, bronchiectasis or active lung infection.
16. Use of Xolair (omalizumab - anti-IgE monoclonal antibody) for 6 months.
17. Immunotherapy with cat or dust mite extract now or in the past.
18. Non-English speakers.
19. History of coagulopathy, thrombocytopenia, pulmonary hypertension, and/or use of anti-coagulants/anti-platelet drugs.

B. Healthy Normal Control Subjects (NC subjects)

Normal control subjects will be individuals who are in good overall health, age and sex matched to the asthmatic group, age 18 - 50 and nonallergic, i.e. entirely negative on the panel of prick skin tests listed in section V (Study Procedures), with no history of allergic rhinitis or asthma, no history of allergic symptoms caused by cats or dust mite allergen exposure, life-long nonsmokers of cigarettes (defined as a lifetime total of less than 5 pack-years and none in 5 years), normal spirometry (i.e. FEV1 and FVC of at least 90% of predicted) and with a methacholine PC20 of > 16 mg/ml.

Exclusion Criteria:

1. A history of allergy, asthma, nasal or sinus disease.
2. Exclusion criteria #1, 3-8 and 10-19 from (A.) above.

C. Allergic Nonasthmatic Subjects (ANA subjects)

Inclusion Criteria:

1. ANA subjects will have a history of either (a) allergic rhinitis (with one or more of the following symptoms: nasal congestion, sneezing, runny nose, postnasal drainage), (b) allergic conjunctivitis (ocular itching, tearing and/or swelling) or (c) contact allergy associated with cat dander or dust mite and a positive allergy test to the same allergen.
2. All subjects will have a baseline FEV1 and FVC determined at the characterization visit that is no less than 90 % of the predicted value.
3. All subjects will have a positive allergy skin prick test to cat dander or dust mite allergen.
4. All subjects will be in good general health.
5. Life-long absence of cigarette smoking (defined as a lifetime total of less than 5 pack-years and none in 5 years).
6. Willing and able to give informed consent.
7. Expressed the desire to participate in an interview with the principal investigator.
8. Age between 18 and 50 years.

Exclusion Criteria:

1. A history of asthma.
2. Exclusion criteria #1, 3-8 and 10-19 from (A.) above.
3. A methacholine PC20 < 16 mg/ml.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 313 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
airway inflammation | 1,6, or 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Medoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Summary and recommendations of a workshop on the investigative use of fiberoptic bronchoscopy and bronchoalveolar lavage in asthmatics. Am Rev Respir Dis. 1985 Jul;132(1):180-2. doi: 10.1164/arrd.1985.132.1.180. PMID 4014864
- [Background] Busse WW, Lemanske RF Jr. Asthma. N Engl J Med. 2001 Feb 1;344(5):350-62. doi: 10.1056/NEJM200102013440507. No abstract available. PMID 11172168
- [Background] Djukanovic R, Wilson JW, Lai CK, Holgate ST, Howarth PH. The safety aspects of fiberoptic bronchoscopy, bronchoalveolar lavage, and endobronchial biopsy in asthma. Am Rev Respir Dis. 1991 Apr;143(4 Pt 1):772-7. doi: 10.1164/ajrccm/143.4_Pt_1.772. PMID 2008989
- [Background] Jarjour NN, Peters SP, Djukanovic R, Calhoun WJ. Investigative use of bronchoscopy in asthma. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):692-7. doi: 10.1164/ajrccm.157.3.9705020. PMID 9517577
- [Background] Kay AB. Allergy and allergic diseases. Second of two parts. N Engl J Med. 2001 Jan 11;344(2):109-13. doi: 10.1056/NEJM200101113440206. No abstract available. PMID 11150362
- [Background] Mackay CR. Chemokines: immunology's high impact factors. Nat Immunol. 2001 Feb;2(2):95-101. doi: 10.1038/84298. PMID 11175800